CLINICAL TRIAL: NCT03031743
Title: Nested Case-control Analysis of the Influence of the Microbiome on Rotavirus Vaccine Immunogenic Response in Infants in Karachi, Pakistan
Brief Title: The Influence of the Microbiome on Rotavirus Vaccine Immunogenic Response in Infants in Karachi, Pakistan
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Aga Khan University (Other); Wageningen University (Other); University of Padova (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Vanessa Harris, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: AIGHD-CSP2013-001
Record Dates: First submitted 2016-07-12; First posted 2017-01-26 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Rotavirus
Keywords: rotavirus vaccine; human microbiome; fecal microbiome; vaccine immunogenicity; Rotarix; immune response, mucosal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- rotavirus (Rotarix TM) vaccination: Infants who received rotavirus vaccination (Rotarix TM) at 6 and 10 weeks, 10 and 14 weeks or 6,10, and 14 weeks. This is a nested study and infants received the vaccination in the overarching study: The Immunogenicity of ROtavirus Vaccine Under Different Age Schedules and the Impact of Withholding Breast Feeding around the Time of Vaccination on the Immunogenicity of Rotarix Vaccine (clinicaltrials.gov: NCT01199874)

SUMMARY:
This is a nested case-control study within an ongoing rotavirus vaccine immunogenicity trial in Karachi, Pakistan. The primary study aim is to compare the fecal microbiota composition and diversity of infants who do (control) and do not (case) demonstrate immune seroconversion to rotavirus vaccination. The infants will be matched for vaccination dose, age and breast-feeding practices.

ELIGIBILITY:
Inclusion Criteria:

* Infants already consented and enrolled in the overarching study: Immunogenicity of Rotavirus Vaccine Under Different Age Schedules and the Impact of Withholding Breast Feeding around the Time of Vaccination on the Immunogenicity or Rotarix Vaccine trial (NCT01199874)

Overarching study (NCT01199874)inclusion criteria:

* 6 weeks 0 days to 7 weeks 6 days age at the time of enrollment
* Healthy infant free of chronic or serious medical condition as determined by history and physical exam at time of enrollment
* written informed consent obtained from parents or guardians for overarching study Nested study additional inclusion criteria
* written informed consent obtained from parents or legal guardians for this nested study
* availability of a baseline, pre-vaccination fecal sample

Exclusion Criteria:

Overarching study (NCT01199874)exclusion criteria

* hypersensitivity to any of the vaccine components
* Use of any investigational drug or vaccine other than the study vaccine within 30 days of first dose of study vaccine or during the study
* use of any immunosuppressive drugs
* previous intussusceptions or abdominal surgery
* enrollment in any other trials
* birth weight less than 1500 grams; or if birthweight is unknown, weight less than 2000 grams on or before 28 days
* immunoglobulin and/or blood products use since birth or during the study period Nested study additional exclusion criteria
* positive serum anti-rotavirus IgA (> or= 20U/mL) at 6 weeks of age, indicative of rotavirus infection prior to vaccination

Ages: 6 Weeks to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants living in a peri-urban slum outside of Karachi, Pakistan
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
differences in fecal microbiota composition | 2 years
  The primary study objective is to see if there are significant differences in the fecal microbiota composition between rotavirus vaccine (Rotarix TM) immune responders (defined as anti-RV IgA antibodies at a concentration of > or = to 20 U/ml in a previously seronegative individual 4 weeks after the last Rotarix dose) and rotavirus vaccine immune non-responders (defined as anti-RV IgA antibodies at a concentration of <20 U/mL 4 weeks after the last Rotarix dose)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa C Harris, MD, Principal Investigator — Amsterdam Institute for Global Health and Development; Academic Medical Center, Amsterdam
Locations (1):
- Aga Khan University, Karachi, Pakistan